CLINICAL TRIAL: NCT05308238
Title: Pre-Active PD: a Randomized Control Trial (RCT) Pilot Study to Improve Self-management of Physical Activity (PA) Routines in Adults with Early-stage Parkinson's Disease (PD)
Brief Title: Pre-Active PD: Looking At Physical Activity Behavior Change in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Jose State University (Other)
Collaborators: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MJF.AOTF.1
Record Dates: First submitted 2022-02-08; First posted 2022-04-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: behavior change; exercise; physical activity; occupational therapy
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled feasibility study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Occupational therapy intervention group (Experimental): Participants will receive 6 telehealth coaching sessions and 8 brief email or text check-ins over the course of 4 months. Participants will also receive a Fitbit and Engage PD Workbook.
  Interventions: Behavioral: Occupational therapy intervention group
- Disease management education group (Active Comparator): Participants will receive online educational videos that they can watch at their own convenience over the course of 4 months. There will be up to 6 hours of content, and the links to these online videos will be provided via email. Following completion of the study, individuals in this group will receive an Engage PD Workbook and one OT coaching session, if they choose to.
  Interventions: Behavioral: Disease management education group

INTERVENTIONS:
Behavioral: Occupational therapy intervention group — Participants will receive 6 telehealth coaching sessions and 8 brief email or text check-ins over the course of 4 months. Participants will also receive a Fitbit and Engage PD Workbook.
  Arms: Occupational therapy intervention group
Behavioral: Disease management education group — Participants will receive online educational videos that they can watch at their own convenience over the course of 4 months. There will be up to 6 hours of content, and the links to these online videos will be provided via email. Following completion of the study, individuals in this group will receive an Engage PD Workbook and one OT coaching session, if they choose to.
  Arms: Disease management education group

SUMMARY:
Pre-Active PD is a randomized controlled feasibility study to evaluate the implementation of a telehealth-delivered physical activity behavior change intervention for people with early-mid stage Parkinson's disease. The program utilizes occupational therapists to provide one-to-one individualized support to facilitate and optimize exercise uptake as part of their disease self-management. The structure of the intervention is based on previous research in neurodegenerative disease including Parkinson's disease and Huntington's disease.

DETAILED DESCRIPTION:
This study will utilize a randomized controlled trial design to assess the feasibility and acceptability of the Pre-Active PD intervention for people with Parkinson's Disease who are in the early disease stage (Hoehn & Yahr stage I or II). The study will compare an experimental group (occupational therapy for exercise behavior change) to a control group (education only). Both groups will be matched for contact time. Individuals will be recruited through the Columbia University Medical Center Parkinson's Disease Center of Excellence. The study will also be listed on the Fox Trial Finder, a website maintained through the Michael J Fox Foundation. Individuals who choose to participate will be screened for eligibility using the inclusion/exclusion criteria and complete the PAR-Q+ safety screen or have medical clearance from their general practitioner. After randomization, participants will be assessed for cognition and history of occupational therapy (OT) and physical therapy (PT). Measures of acceptability will include retention and completion rates, Fitbit wear-time, and the Perceived Autonomy Support Healthcare Climate Questionnaire (PAS-HCCQ). Implementation will be assessed by the Rating Tool to Assess Fidelity of Intervention Delivery. Physical activity levels will be measured by a wearable activity monitor (Actigraph™ GT9X), worn 7 consecutive days pre and post intervention and 2nd follow-up, as well as a questionnaire. We will also use the Self-Efficacy for Exercise Scale and measure balance and mobility. Descriptive statistics (mean, standard deviation) will be calculated for all demographic information and resultant outcome measures.

Baseline and follow-up outcome measures include the following domains: exercise self-efficacy scale, exercise motivation (Behavioral Regulation In Exercise Questionnaire, physical activity levels (Brunel Lifestyle Physical Activity Questionnaire; ActiGraphTM wearable activity monitor, and Modified PA-R Question), physical performance measures (TUG Single Task and Dual Task Cognitive Version; 30 second sit-to-stand; Modified 2 Minute Step Test), self-perception measures (Modified Canadian Occupational Performance Measure; Patients' Global Impression of Change scale), and the Life Space Assessment.

Participants assigned to the occupational therapy intervention group, will receive 6 telehealth coaching sessions and 8 brief email or text check-ins over the course of 4 months. They will also receive a Fitbit and Engage PD Workbook. The third coaching session will be audio and video-recorded (if consented) and later viewed by an assessor to determine how well the intervention was delivered. The recording will be stored until completion of the study. Declining to be recorded will not affect study participation.

The OT intervention group will utilize the Pre-Active PD program (Clinicaltrials.gov NCT03696589) to guide the delivery of the intervention. This will include a checklist of the key elements that are important for the therapist in order to facilitate PA behavior change. In addition, the therapist will utilize motivational interviewing strategies that include four processes (engaging, evoking, planning, and tracking) and five core communication skills (asking open ended questions, affirming, reflective listening, summarizing, and informing and advising). The therapist will introduce the Pre-Active PD workbook and utilize it as a tool and reference for the participant in order to engage and focus them throughout the coaching process, and will educate participants on the types of exercise options and the specific exercise benefits for PD. In the planning process, the therapist will facilitate discussion on development of specific and measurable goals, and will give the participant a Fitbit physical activity monitor so that they can self-monitor their heart rate and physical activity during the course of the intervention period. The recommended exercises will be individualized to each participant but will primarily focus on increasing general physical activity (e.g. steps per day) as well as engagement in moderate-vigorous intensity aerobic exercise a minimum of three times per week. Balance and strengthening exercises will also be recommended as appropriate. Participants will also be given a short exercise safety checklist to assure safety when conducting home exercises.

Participants assigned to the disease management education group, will receive online educational videos that can be watched at their own convenience over the course of 4 months. There will be up to 6 hours of content, and the links to these online videos will be provided via email. Following completion of the study, individuals in the control group will receive an Engage PD Workbook and one OT coaching session.

ELIGIBILITY:
Inclusion Criteria:

1. Neurologist confirmed clinical dx for Parkinson's disease Hoehn & Yahr stage I or II
2. Ambulatory for indoor and outdoor mobility without assistance or assistive device
3. Successful completion of Physical Activity Readiness Questionnaire (PAR-Q), or medical clearance from GP

Exclusion Criteria:

1. Musculoskeletal injury that would prevent participation in an exercise program
2. Other neurological diseases or disorders such as stroke
3. Already engaging in aerobic exercise for at least 30 minutes for 5 or more days per week.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Feasibility: Adherence | 4 months
  Participant completion of ≥ 75% of sessions 1, 2 & 3
Feasibility: Retention | 4 months
  > 75% of all participants retained at follow-up
Change from baseline Brunel Lifestyle Physical Activity Questionnaire (Karageorghis, 2005) at 4 months and 6 months | Baseline, 4 months, and 6 months
  A 10-item questionnaire that measures both pre-planned (6 items) and un-planned (3 items) lifestyle PA. Scoring for each item is on a scale of 1-5, and the scores for each subscale are averaged. Scores range from 1 (low level of physical activity) to 5 (high level of physical activity).
Change From Baseline Moderate-Vigorous Physical Activity Using Actigraph at 4 Months and 6 months | Baseline, 4 months, and 6 months
  Measured using ActiGraph accelerometer, levels of moderate-vigorous physical activity will be measured, as well as number of steps and sedentary behavior.

SECONDARY OUTCOMES:
Change From Baseline Timed-up-and-go (TUG) at 4 Months and 6 months | Baseline, 4 months, and 6 months
  Participant starts sitting in chair and then rises when prompted to "go" and then walks 3 meters, turns around, walks back to chair and sits. Time to complete is recorded. Then it is performed again with the additional element of counting backwards by 3 starting at a randomly selected number between 20 and 100.
Change From Baseline 30 second sit-to-stand at 4 Months and 6 months | Baseline, 4 months, and 6 months
  A physical performance measure which assesses functional lower extremity strength in older adults. The person is seated in a chair without arms, with feet shoulder width apart (placed on floor), and arms crossed over the chest. The participant is then encouraged to complete as many full stands as possible within 30 seconds. The number of full stands completed with the 30 sec period is the score.
Change From Baseline Modified 2 Minute Step Test at 4 Months and 6 months | Baseline, 4 months, and 6 months
  A physical performance assessment to determine a participant's cardiorespiratory fitness level. This will be completed with a caregiver (virtually trained on proper guarding) present to ensure safety.
Change From Baseline Perceived Functional Ability (PFA) Questionnaire (George et al., 1997) at 4 Months and 6 months | Baseline, 4 months, and 6 months
  2-question assessment that quantifies participants' perceived ability to complete a 1- and 3-mile distance at a comfortable pace from a scale of 1 (slow-pace) to 13 (fast pace)
Change From Baseline Modified Canadian Occupational Performance Measure (Dedding et al., 2004) at 4 Months and 6 months | Baseline, 4 months, and 6 months
  This is a questionnaire used to determine participant goals and allows participants to rate current satisfaction, importance, and performance on these goals. A scale of 1 (not satisfied at all) to 10 (extremely satisfied) is used.
Change From Baseline Patients' Global Impression of Change scale (Hurst & Bolton, 2004) at 4 Months | Baseline, and 4 months
  Self-perception of change
Change From Baseline Life Space Assessment (Stalvey et al., 1999) at 4 Months and 6 months | 0, 4 & 6 months
  Questionnaire that determines how much the person gets out and about and the spatial extent of the person's typical life space, i.e., what is the usual range of places in which the person engages in activities within the designated time frame.
Post-Intervention Acceptability Questionnaire | 4 months
  Structured questionnaire based on Theoretical framework of acceptability (TFA)
Intervention Implementation | 4 months
  Rating Tool to Assess Fidelity of Intervention Delivery (Quinn, Trubey, et al., 2016)
Change From Baseline Modified PA-R Questionnaire at 4 Months | 0 & 4 months
  1-question self-rating of physical activity level over past 6-months.
Perceived Autonomy Support Healthcare Climate Questionnaire (HCCQ) (Williams, Freedman, & Deci, 1998): | 4 months
  A short questionnaire to assess intervention acceptability

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Jose State Universty, San Jose, California
  - Neurorehabilitation Research Laboratory, New York, New York

IPD SHARING:
Plan to Share IPD: No